CLINICAL TRIAL: NCT06296823
Title: Biomarkers for Peripheral Circadian Clocks in Humans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Kenneth Wright, Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 22-0466
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Circadian Rhythms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meal timing (Experimental): Three days of meals, bedtimes and wake times scheduled to occur 5h earlier.
  Interventions: Behavioral: Simulated jetlag protocol
- Bright light (Experimental): Three days of exposure to bright light of ~3,000 lux, which is less than one-third the brightness of a sunrise or sunset (timed to start earlier by 1h each day) with scheduled bed and wake times timed 5h earlier.
  Interventions: Behavioral: Simulated jetlag protocol

INTERVENTIONS:
Behavioral: Simulated jetlag protocol — 16 hours of wakefulness and an 8 hour scheduled sleep opportunity in a simulated jetlag protocol where you will go to bed and awaken earlier than usual.

SUMMARY:
The purpose of this project is to improve our understanding of peripheral circadian rhythms in humans. Circadian clocks are present in most tissues of the body with importance for optimal physiological function, health, and behavior. This project will utilize simulated jetlag protocols to systematically test novel hypotheses about the regulation of peripheral circadian rhythms in humans. Specifically, we will examine how changes in the time of when we are exposed to light and the timing of when we eat impacts proteins in the blood and saliva that represent rhythms from clocks in the brain (e.g., rhythms of the hormones melatonin and cortisol coordinated by the brain) and rhythms from clocks in body tissues (e.g., proteins made by immune and bone cells, and cells in the stomach and liver). We also aim to discover new blood-based biomarkers of peripheral rhythms in humans. We anticipate our findings will be the first step in developing novel circadian based treatments for aligning peripheral clocks under conditions such as jetlag, and for developing novel circadian biomarkers that will advance our scientific understanding of circadian rhythms.

DETAILED DESCRIPTION:
Visit 1: Participants who meet pre-screen/initial inclusion criteria will be consented at Visit 1, complete additional questionnaires and interviews to assess inclusion/exclusion criteria, and we will collect descriptive data as well as have our clinical psychologist perform a clinical interview.

Visit 2: Participants will undergo medical screening at the Clinical Translational Research Center at the University of Colorado Boulder (UCB-CTRC) to determine health status.

Visits 3 & 6: Participants will be asked to maintain a regular ~8h sleep-wake schedule for two weeks prior to Visits 5 and 8. Participants will wear a wrist activity, skin temperature, and light exposure recorder. Participants will be asked to remain in the local time zone during ambulatory recording procedures and be asked to keep their typical schedules (e.g., not stay up all night for work or social events and not reside in a new place different from their place of residence).

Visit 4 & 7: Participants will come to the laboratory on days 11 and 39, where qualified staff will apply a Continuous Glucose Monitoring (CGM) sensor to be worn for ~3 days at home and will continue in the laboratory. For the three days leading up to the study isocaloric meals including breakfast, lunch, and dinner will be provided. Participants will be asked to consume these energy balanced research diets (no caffeine) and meal timing will be scheduled (breakfast ~30 min, lunch ~5h, and dinner ~10h after awakening,). Exercise will be proscribed for these 3-days prior to the in-lab study.

Visits 5 & 8: Participants will be randomized to condition order using an ABBA design (i.e., randomized into one of the two experimental conditions first in a crossover design: 3-days bright light exposure or 3-days of earlier timed meals). Both conditions are tested under an advanced sleep-wake schedule equivalent to traveling 5 time zones east. All participants will complete both conditions. On the second visit, participants will be tested in the other condition. Participants will live in the laboratory for 7.7 days each visit.

ELIGIBILITY:
Inclusion Criteria:

1) 17-35 years old 2) English speaking 3) Healthy 5) Altitude history: Currently residing at Denver altitude or higher

Exclusion Criteria:

1. Any medical, psychiatric, or sleep disorder.

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
PYY | hourly for up to 25 hours on two occasions
  Appetitive hormone-promotes satiety
Ghrelin | hourly for up to 25 hours on two occasions
  Appetitive hormone-promotes food intake
Leptin | hourly for up to 25 hours on two occasions
  Appetitive hormone-promotes satiety
CRP | hourly for up to 25 hours on two occasions
  Acute phase response/also marker of inflammation
OMD | hourly for up to 25 hours on two occasions
  Biomineralization
PAI-1 | hourly for up to 25 hours on two occasions
  Inhibitor of fibrinolysis
IgE | hourly for up to 25 hours on two occasions
  Immune responses to parasites and allergens
CCL18 | hourly for up to 25 hours on two occasions
  Chemotaxis / immune cell trafficking
PTH | hourly for up to 25 hours on two occasions
  Serum calcium homeostasis

SECONDARY OUTCOMES:
Glucose | continuously for up to 35 hours on two occasions
  Blood sugar
Insulin | hourly for up to 25 hours on two occasions
  hormone that helps regulated blood glucose levels
Proteomics | hourly for up to 25 hours on two occasions
  proteins

OTHER OUTCOMES:
Melatonin | hourly for up to 25 hours on two occasions
  Primary marker of the SCN master clock - high levels represent biological night
Cortisol | hourly for up to 25 hours on two occasions
  Secondary marker of the SCN master clock - rising/high levels represent biological night
Core body temperature | continuously for up to 35 hours on two occasions
  Secondary marker of the SCN master clock - low levels represent biological night
Skin temperature | continuously for up to 35 hours on two occasions
  Secondary marker of the SCN master clock - high levels represent biological night
Cognition | hourly for up to 35 hours on two occasions
  Measures of performance
Blood pressure | hourly for up to 35 hours on two occasions
  systolic and diastolic pressures
Metabolomics (grant application planned to analyze not currently funded) | hourly for up to 25 hours on two occasions
  small molecules in the plasma
Oral microbiome (grant application planned to analyze not currently funded) | hourly for up to 25 hours on two occasions
  oral bacteria
Skin microbiome (grant application planned to analyze not currently funded) | hourly for up to 25 hours on two occasions
  skin bacteria

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep and Chronobiology Laboratory, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Any data generated from the proposed work that is presented in a peer reviewed journal will be de-identified.
  Other data that is presented in a peer reviewed journal will be archived indefinitely and made available upon request.
  Microbiome data will be deposited in the International Nucleotide Sequence Database Collaboration www.insdc.org/ and is already deposited in Qiita http://qiita.microbio.me
  Metabolomics data will be deposited in Global Natural Products Social (GNPS) molecular networking http://gnps.ucsd.edu
Time Frame: Upon publication, microbiome data to be deposited permanently in International Nucleotide Sequence Database Collaboration www.insdc.org/ Data deposited in Qiita http://qiita.microbio.me Upon publication, proteomics and metabolomics data to be deposited and made freely available (e.g., https://figshare.com, http://gnps.ucsd.edu)
Access Criteria: microbiome, proteomics and metabolomics data will be freely available at www.insdc.org/, https://figshare.com, and http://gnps.ucsd.edu